CLINICAL TRIAL: NCT05122520
Title: A Questionnaire to Identify Predictive Symptoms and Risk Factors for Hydrogen and Methane Breath Testing Outcomes
Brief Title: Hydrogen and Methane Breath Test Questionnaire
Acronym: HMBTQ
Status: Completed | Type: Observational
Sponsor: The Functional Gut Clinic (Other)
Responsible Party: Principal Investigator, Dr Anthony Hobson, Clinical Director, The Functional Gut Clinic
Other Study IDs: FGC-20-003
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Small Intestinal Bacterial Overgrowth
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The HMBT-Q is a 26-item questionnaire, split into four main sections: food related symptoms; general digestive symptoms; extra-intestinal symptoms and co-morbidities and Medication and onset.

SUMMARY:
Lactulose HMBT and Glucose HMBT are simple non-invasive tests to assess whether imbalances in gut bacteria may be contributing to troublesome tummy symptoms. These imbalances in gut bacteria include small intestinal bacterial overgrowth (SIBO) and excessive methane production.

Recently there has been a lot of work to done by experts in the field, to ensure that performance and interpretation of these tests are standardised, to help improve the clinical utility of these investigations. Although there is a lot of information currently available demonstrating the risk factors and symptoms associated with these conditions, there is a lack of data demonstrating the factors that might lead to a positive test according to these new parameters. This study aims to collect data on symptoms and medical history, in patients referred for lactulose and glucose HMBT in order further improve the effectiveness of this test in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is referred for and able to complete a postal Lactulose or Glucose HMBT according to protocol with The Functional Gut Clinic
2. Participant has capacity to understand written English
3. Participant can communicate well with the Investigator and to comply with the requirements for the entire study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients referred for Glucose and Lactulose HMBT at the Functional Gut Clinic will be approached to see if they would like to take part in this study
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Determine positive predictive symptoms for SIBO positive participants determined by HMBT | At same time as breath test
  Using the HMBTQ

SECONDARY OUTCOMES:
Determine positive predictive symptoms for excessive methane positive participants determined by HMBT | At same time as the breath test
  Using the HMBTQ
Determine the frequency of recognised and potential risk factors in SIBO positive participants | At the same time as the breath test
  Using the HMBTQ
Determine the frequency of recognised and potential risk factors in excessive methane positive participants | At the same time as the breath test
  Using the HMBTQ

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hobson, Principal Investigator — The Functional Gut Clinic
Locations (1):
- The Functional Gut Clinic, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided